CLINICAL TRIAL: NCT02245724
Title: Stem Cell Therapy in Mental Retardation
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Neurogen Brain and Spine Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NGBSI-15
Record Dates: First submitted 2014-09-12; First posted 2014-09-22 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Mental Retardation
Keywords: Mental retardation; Autologous mononuclear cell therapy; Stem cell
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stem Cell (Experimental): Bone marrow mononuclear cell transplantation
  Interventions: Biological: Stem Cell

INTERVENTIONS:
Biological: Stem Cell — Autologous bone marrow mononuclear cell transplantation

SUMMARY:
The purpose of this study was to analyze the benefit of autologous mononuclear cell therapy in mental retardation.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed cases of mental retardation
* age above 6 months

Exclusion Criteria:

* presence of acute infections such as Human immunodeficiency virus/Hepatitis B Virus/Hepatitis C Virus
* malignancies
* bleeding tendencies
* pneumonia
* renal failure
* severe liver dysfunction
* severe anemia [Hemoglobin < 8]
* any bone marrow disorder
* space occupying lesion in brain
* other acute medical conditions such as respiratory infection and pyrexia

Ages: 6 Months to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2011-09; Primary Completion 2016-03 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change in common clinical symptoms of mental retardation | 1 year
  Change in symptoms such as cognition, remote memory, problem solving,understanding of relationships,social interaction,communication,self care, activities of daily living will be recorded at 1 year follow up.

CONTACTS AND LOCATIONS:
Locations (1):
- Neurogen brain and spine institute, Navi Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sharma A, Sane H, Gokulchandran N, Pai S, Kulkarni P, Ganwir V, Maheshwari M, Sharma R, Raichur M, Nivins S, Badhe P. An open-label proof-of-concept study of intrathecal autologous bone marrow mononuclear cell transplantation in intellectual disability. Stem Cell Res Ther. 2018 Jan 31;9(1):19. doi: 10.1186/s13287-017-0748-2. PMID 29386049